CLINICAL TRIAL: NCT00338507
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter, Placebo-Controlled Dose_Ranging Study of Erdosteine for the Treatment of Stable Chronic Bronchitis Associated With Chronic Obstructive Pulmonary Disease
Brief Title: Phase 2 Study - Erdosteine in Patients With CB/COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adams Respiratory Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERD-CB-01-2005
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Chronic Bronchitis; Chronic Obstructive Pulmonary Disease
Keywords: Chronic Bronchitis; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive | interventions — erdosteine

INTERVENTIONS:
Drug: Erdosteine

SUMMARY:
This clinical study is designed to explore dose ranging and identify methods to demonstrate the efficacy of Erdosteine in patients with stable Chronic Bronchitis associated with Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a clinical diagnosis of stable CB associated with COPD will be entered into this study. CB is diagnosed clinically in patients who have a documented smoking history and who have a daily productive cough for at least 3 months per year over at least 2 consecutive years in the absence of other causes of chronic cough. COPD is defined by the presence of airflow obstruction from spirometry

Exclusion Criteria:

asthma, bronchiectasis, or cystic fibrosis; active history of lung cancer, respiratory failure, or a need for long-term oxygen therapy;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Albrecht, MD, Study Director — Adams Respiratory Therapeutics
Locations (1):
- Omnicare Clinical Research, King of Prussia, Pennsylvania, United States